CLINICAL TRIAL: NCT06218836
Title: Effect of Kinetic Contact-friction Modulation With a Pre-inflated Tracheal Tube Cuff on Postoperative Sore Throat in Adults With Anticipated Non-difficult Airway: a Randomized Controlled Study
Brief Title: Effect of Inflated Versus Non-inflated Endotracheal Tube on Sore Throat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/12/23/2408
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Sore Throat
Keywords: endotracheal tube; inflated; sore throat; friction
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into two groups:
  Group I: Intubation with pre-inflated endotracheal tube Group II: Intubation with non-inflated endotracheal tube
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent investigator, not involved in the assessment of patient, will assign the allocated intervention. The patient and the postoperative outcome assessor will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubation with pre-inflated ETT (Active Comparator): Patient's trachea will be intubated using pre- inflated endotracheal tube (ETT)
  Interventions: Other: Pre-inflated endotracheal tube
- Intubation with non-inflated ETT (Active Comparator): Patient's trachea will be intubated using non-inflated ETT
  Interventions: Other: Non-inflated endotracheal tube

INTERVENTIONS:
Other: Pre-inflated endotracheal tube — The ETT (males: size 7.5 mm ID, females: size 6.5 mmID) will be taken out from the wrapper and submerged in 0.9% normal saline till the proximal margin of the cuff. Then, the cuff will be inflated to 40 cm of H2O to gain full stretch inflation.Thereafter the cuff will be deflated with the help of cuff inflator-deflator device to maintain intracuff pressure of 4 cm H2O The external cuff balloon will be obliterated with a soft clamp to ensure that at the time of passage of tube through the glottic-inlet, the tube cuff does not get deflated due to pressure equalization with the external balloon.
  Arms: Intubation with pre-inflated ETT
Other: Non-inflated endotracheal tube — The ETT (males: size 7.5 mm ID, females: size 6.5 mmID) will be taken out from the wrapper and submerged in 0.9% normal saline till the proximal margin of the cuff. Thereafter the endotracheal intubation will be done.
  Arms: Intubation with non-inflated ETT

SUMMARY:
Postoperative sore throat (POST) is a common morbidity following upper airway access-control with direct laryngoscopy-intubation (DLI) technique. Various reasons (size of the tracheal tube, cuff pressure, rough tube pass, and reattempts, among others) have been cited and management strategies (pharmacologic: applying lidocaine gel/EMLA cream on the cuff surface; non-pharmacologic measures: tracheal tube cuff pressure control, optimization of tracheal tube size, applying lubricating gel) have been tried, but none has been able to decrease the incidence of POST nor has been able to decrease the suffering of patients.

Traditionally, intubation is performed with a deflated endotracheal tube and the cuff is later inflated to secure the tube in desired position. The striated folds present in the deflated cuff incurs additional dynamic friction that traumatizes upper airway mucosa during the procedure, causing the risk of POST. While accentuated friction burden on the posterior part of vocal cords and the tracheal mucosa has been studied recently, there has been no work on understanding the kinetic contact- friction ensued by a passing tracheal tube/cuff. We speculate that dynamic contact-friction generated at the time of passing of a cuffed tracheal tube is the major active component which has potential to cause actual tissue trauma and inflammation resulting in adverse effects (POST, hoarseness, throat pain, cough). This study aims to evaluate the effects of reducing dynamic/kinetic contact-friction by employing a pre-inflated tracheal tube cuff to pass the vocal cords at the time of orotracheal intubation.

DETAILED DESCRIPTION:
Postoperative sore throat (POST) has long been a common and nagging complication following conventional direct laryngoscopy-intubation (DLI) procedure. A significant quantum of POST incidence during DLI in non-difficult airway (NDA) could be attributed to inter-operator variability in approach, experience, proficiency, and equipment (e.g., type of laryngoscope/tracheal tube). Additional factors determining the occurrence of POST, include size of the tracheal tube, cuff pressure, rough tube pass, and reattempts, among others. Several pharmacologic (applying lidocaine gel, inhaled corticosteroids and EMLA cream on tracheal tube cuff surface) and non- pharmacologic measures/modalities (e.g., tracheal tube cuff pressure control, optimization of tracheal tube size, applying gel) have been employed to preclude/diminish POST, however, neither the incidence nor the suffering of patients have come down yet following these interventions. Friction injury to the tracheal mucosa during the passage of ETT is one of the important contributing factors to POST but has not been adequately evaluated. Friction injury to the upper airway mucosa not only occurs during rough or repeated passage of ETT through the glottic-inlet but also when the ETT cuff comes in contact with the tracheal mucosa during dynamic passage of ETT through the glottis.

Traditional approach to reduce reduce postoperative sore throat is by containing the intracuff pressure with use of non-inflated tube, and consequently, reducing static pressure burden on tracheal mucosa. No study has explored the impact of modulation of obligate kinetic contact-friction that occurs during passage of tube across the glottic-inlet. A preemptive limited inflation of tracheal tube cuff before actual intubation may modulate the kinetic-contact friction during the passage of the tracheal tube cuff past the vocal cords, and hence may help reduce postoperative sore throat in these patients. We plan this randomized trial to compare the effect/efficacy of intubation with pre-inflated tracheal tube on the incidence of postoperative sore throat in patients with anticipated non-difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* Patients with anticipated non-difficult airway with the following characteristics:

  i. Normal head and neck movements ii. Adequate mouth opening iii. No retrognathia or prognathia iv. Normal dentition
* Surgeries with anticipated duration of 40 minutes - 3 hours

Exclusion Criteria:

* Obese patients (BMI > 33 kg/m2)
* Requiring use of intubation aids such as bougie, stylet or video-laryngoscope
* Recent history of steroid or non-steroidal anti-inflammatory drug use
* Systemic illness with presenting complaints of sore/dry throat (diabetics with polydipsia, hypertensives on diuretics, moribund bed ridden patients)
* History of airway related morbidity post operative sore throat [POST]
* Patients with a history of chronic smoking (1 pack per day for 10 years) chewing tobacco, and tobacco-related products
* Patients undergoing head and neck, intraoral/nasal surgery, or recent history of such surgery
* Patients with a past surgical history of tracheostomy (post decannulation)
* Surgery in prone position
* Ongoing upper and lower respiratory tract inflammation/infection
* Patients with anticipated postoperative mechanical ventilation
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat | From time of extubation of trachea till 24-hours postoperatively
  Sore throat will be assessed using a 4-point scale: '0' no sore throat to '3' severe sore throat.Any score >= 1 will be counted as a sore throat incidence

SECONDARY OUTCOMES:
Severity of postoperative sore throat | From time of extubation of trachea till 24-hours postoperatively
  Sore throat will be assessed using a 4-point scale: '0' no sore throat, '1' Mild sore throat (complained of sore throat only on enquiry), '2' Moderate sore throat (complained of sore throat on his/her own), and '3' Severe sore throat (change of voice or hoarseness). Number of patients with no sore throat, mild sore throat, moderate sore throat, and severe sore throat will be noted
Incidence and severity of postoperative cough | From time of extubation of trachea till 24-hours postoperatively
  Postoperative cough will be assessed using a 4-point scale: 0- no cough, 1- mild cough (cough which is less than a common cold), 2-moderate cough (cough which is similar to a common cold), and 3- severe cough (cough which is more than a common cold).
Incidence and severity of postoperative hoarseness of voice | From time of extubation of trachea till 24-hours postoperatively
  Postoperative hoarseness of voice will be assessed using a 4-point scale: 0- no hoarseness (no change in speech appreciated even on enquiry), 1- mild hoarseness (minimal change in speech quality. Answered by patient on enquiry), 2-moderate hoarseness (moderate change in speech quality which is self-complained by the patient), and 3- severe hoarseness (recognizable change in speech quality).

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dutta, MD, PGDHR, Study Director — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No